CLINICAL TRIAL: NCT00176280
Title: A Randomized Phase II Trial of Pre-chemotherapy Leukine vs. Leukine-Dexamethasone in Combination With Gemcitabine and 5-Fluorouracil (5-FU) in Patients With Metastatic Renal Cell Carcinoma (RCC)
Brief Title: Randomized Phase 2 Trial of Pre-chemotherapy Leukine vs. Leukine-Dexamethasone in Combination With Gemzar & 5-FU in Patients With Metastatic Renal Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Kentucky (Other)
Collaborators: Bayer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-GU-51-B
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal; Carcinoma; Renal Cell Carcinoma; RCC; Leukine; Dexamethasone; Gemcitabine; 5 Fluorouracil; 5 FU; Metastatic
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma; Neoplasm Metastasis | interventions — sargramostim; Dexamethasone

INTERVENTIONS:
Drug: Leukine
Drug: Dexamethasone

SUMMARY:
-Overall study design: A randomized Phase II study in patients with metastatic RCC Patients will receive chemotherapy with gemcitabine and 5-FU. Prior to each chemotherapy the patient will receive a combination of Leukine alone (study cohort 1) or Leukine-dexamethasone (study cohort 2).

-Chemotherapy: gemcitabine 1.0 g/m2 intravenously (infused in the vein)over 30 minutes on Days 7 and 21, Folinic acid 200 mg/m2 on Days 7-8 and 21-22, then 5-FU 400 mg/m2, intravenously (infused in the vein) over 30 minutes followed by 5-FU 600 mg/m2 intravenously (infused in the vein) over 24 hours.

•Study drugs:

* Cohort 1, Leukine, 250 ug/m2 daily (8 am) subcutaneously (under the skin) on days 1, 2, 3, 4, 5 and 15, 16, 17, 18, and 19;
* Cohort 2, Leukine, 250 ug/m2 daily (8 am) subcutaneously (under the skin)on days 1, 2, 3, 4, 5, and 15, 16, 17, 18, and 19 and dexamethasone 12 mg every 12 hours (8 am and 8 pm) orally (by mouth) on days 3, 4, 5, 6, 7, 17, 18, 19, 20, and 21.

DETAILED DESCRIPTION:
STUDY SYNOPSIS

Objectives:

Primary:

1. Determine the response rates and overall survival in patients with metastatic renal cell carcinoma (RCC) receiving pre-treatment with Leukine-dexamethasone vs Leukine alone in combination with gemcitabine-5-FU.
2. Determine if pre-treatment with the combination of Leukine-dexamethasone is more effective than pre-treatment with Leukine alone in reducing the hematopoietic and non-hematopoietic toxicities of gemcitabine-5-FU in patients with metastatic RCC.

Secondary:

1. Determine the effects of the combination of Leukine-dexamethasone vs Leukine alone on the number and function of peripheral blood dendritic cells, and cytokine levels when given prior to gemcitabine-5-FU in patients with metastatic RCC.
2. Determine quality of life and toxicity of treatment in patients with metastatic RCC receiving pre-treatment with Leukine-dexamethasone vs Leukine alone in combination with gemcitabine-5-FU.
3. Determine the dose intensity administered in both treatment groups.

Study Design:

* Overall study design: A randomized Phase II study in patients with metastatic RCC Patients will receive chemotherapy with gemcitabine-5-FU. Patients will receive prior to each chemotherapy the combination of Leukine alone (Cohort 1) or Leukine-dexamethasone (Cohort 2).
* Patient eligibility: a) chemotherapy naive patients with biopsy proven RCC, b) PS (ECOG), 0, 1, or 2, c) measurable disease by RECIST criteria, d) previous immunotherapy and anti-angiogenic therapy is allowed, e) adequate bone marrow, renal and hepatic function as defined by AGC > 1500 and PLC > 100,000 mm3 and serum creatinine and bilirubin < 1.5 mg/dl.
* Chemotherapy: Cohorts 1 and 2: Days 7 and 21: gemcitabine 1.0 g/m2 intravenously over 30 minutes; Days 7-8 and 21-22: Folinic acid 200 mg/ m2, then 5-FU 400 mg/ m2, intravenously over 30 minutes followed by 5-FU 600 mg/ m2 intravenously over 24 hours.
* Study Drugs:

  * Cohort 1, Leukine, 250 ug/m2 daily (8 am) subcutaneously days 1, 2, 3, 4, 5, and 15, 16, 17, 18, and 19;
  * Cohort 2, Leukine, 250 ug/m2 daily (8 am) subcutaneously days 1, 2, 3, 4,5, and 15, 16, 17, 18, and 19 and dexamethasone 12 mg every 12 hours (8 am and 8 pm) orally days 3, 4, 5,6, 7, 17, 18, 19, 20, and 21.
* Evaluations during this trial: Baseline: history and physical examination with vital signs/weight, estimation of performance status (PS), CAT scans of chest, abdomen and pelvis, EKG, CBC/differential, urinalysis, complete biochemistry profile (CMP) (12 component) and quality of life assessment. Prior to each course: interim history, physical examination with vital signs/weight, grading of all toxicities, and estimation of PS, CMP, and CBC/differential. Prior to course 3, 5, and thereafter (every other course): CAT scans of chest, abdomen, and pelvis, tumor response and quality of life assessment. Each week after initiation of study (ie day1, course 1): CBC/differential, x 3 (Monday Wednesday and Friday). Biologic studies to include assessment of dendritic cell number and function (20 ml blood), days 1 and 7 of course 1.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically proven, metastatic RCC. Patients may have either recurrent or primary Stage IV or unresectable regionally advanced disease.
2. Previous surgery (nephrectomy), immunotherapy with IL-2, IFN-a or other cytokines and anti-angiogenic therapy are allowed but all therapy must have been completed four weeks prior to entry into this study.
3. Previous radiation therapy is allowed if completed at least four weeks prior to study entry and therapy was administered to < 25% of the bone marrow.
4. Patients must be >18 years of age (age limit required by the State of Kentucky). Women of childbearing potential must have a negative pregnancy test and must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
5. Patients must have ECOG PS 0,1 or 2.
6. Patients must have at least one target lesion according to the RECIST criteria. Bone metastases, leptomeningeal disease, ascites, pleural or pericardial effusions, lymphangitic spread or cystic lesions are not acceptable as target lesions.
7. Patients must have an expected survival of at least four months.
8. Patients must have adequate organ and marrow function as defined as follows: leukocytes >3,000/mm3, absolute neutrophil count >1,500/mm3, hemoglobin >8.0g/dl, platelets >100,000/mm3, total bilirubin and serum creatinine must be < 1.5 mg/dl. Liver transaminases (SGOT and/or SGPT) may be up to 2.5 institutional upper limit of normal (ULN) if alkaline phosphatase is <ULN or alkaline phosphatase may be up to 4 ULN if transaminases are <ULN.
9. Patients must have the ability to understand and the willingness to sign a written informed consent document. Patients have the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria:

1. Patients with previous history of cancer are excluded unless they have had curative treatment completed >5 years prior to entry onto study or have one of the following: in situ carcinoma (any location), basal cell carcinoma, or non-metastatic squamous cell carcinoma of the skin.
2. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled or untreated cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients requiring any non study corticosteroids for any reason are excluded.
4. Pregnant women are excluded from this study because of the teratogenic potential of 5-FU and gemcitabine. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Lactating women are also excluded. Post menopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
5. Patients may not be receiving any other investigational agents.
6. Peripheral neuropathy must be ≤ grade 1.
7. Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the Investigator to be significant enough to preclude informed consent or interfering with compliance for oral drug intake are excluded.
8. Major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from major surgery.
9. Participation in any investigational drug study within 4 weeks preceding treatment start.
10. Lack of physical integrity of the upper gastrointestinal tract or those who have malabsorption syndrome or inability to swallow tablets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09

PRIMARY OUTCOMES:
% of subjects with CR or PR evaluated after course 2 then every other course using RECIST for both cohorts
Survival (assessed until death)
QOL (evaluated after courses 3 & 5 then every other course)
% of subjects with >/= grade 3 hematopoietic & non-hematopoietic toxicities (assessed 3/week on treatment & continuing until counts recover)

SECONDARY OUTCOMES:
Days with <AGC 500 & platelet (PLC)< 20K mm3, # of febrile neutropenia hospital days, # of transfusions, bleeding & # of outpatient antibiotic days (assessed 3/week on treatment then until counts recover)
Levels of peripheral blood dendritic cell # & function, plasma levels of cytokines including VEGF & TNF alpha (performed on days 1 & 7 of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: John Rinehart, MD, Study Chair — University of Kentucky